CLINICAL TRIAL: NCT03017300
Title: Transdiaphragmatic Pressure and Neural Respiratory Drive Measured During Inspiratory Muscle Training in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Weiliang Wu, PHD, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GuangzhouInRD; GuangzhouIntRD (Other: Guangzhou Institute of Respiratory Disease)
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- COPD（threshold IMT training） (Experimental): COPD patient use Inspiratory muscle trainer (Threshold IMT®)
  Interventions: Device: Threshold IMT®
- COPD（resisive training） (Experimental): COPD patient use Inspiratory muscle trainer (PFLEX®)
  Interventions: Device: PFLEX®

INTERVENTIONS:
Device: Threshold IMT® — A device used to offer threshold load to inspiratory muscle
  Other Names: inspiratory threshold load inspiratory muscle training
  Arms: COPD（threshold IMT training）
Device: PFLEX® — A device used to offer resisive to inspiratory muscle
  Other Names: inspiratory resisive inspiratory muscle training
  Arms: COPD（resisive training）

SUMMARY:
Inspiratory muscle training（IMT）was an rehabilitation therapy for stable patients with chronic obstructive pulmonary disease(COPD). However, its therapeutic effect remains undefined due to unclear of diaphragmatic mobilization during IMT. Diaphragmatic mobilization represented by transdiaphragmatic pressure（Pdi）and neural respiratory drive expressed as corrective root-mean-square(RMS) of diaphragmatic electromyogram(EMGdi) provide vital information to select the proper IMT device and loads in COPD, therefore make curative effect of IMT clarity. Pdi and RMS of diaphragmatic electromyogram (RMSdi%) was respectively measured and compared during inspiratory resistive training and threshold load training in stable patients of COPD.

DETAILED DESCRIPTION:
Subjects：The diagnosis and severity of all participants were measured using the pulmonary function test according to Global Initiative for Chronic Obstructive Lung Disease.

Inclusion criteria: (1)Severe and very severe COPD (postbronchodilator FEV1/FVC under 70% and FEV1 under 50% of the predicted value (GOLD C and D group); (2)Inspiratory muscle weakness（Maximal Inspiratory Pressure under 60cmH2O）; (3) Bronchial dilation test (BDT) negative.

Exclusion criteria: (1) acute exacerbation in the previous 4 weeks; (2) using the oral corticosteroids within4 weeks; (3) history of other respiratory, cardiovascular, neuromuscular, musculoskeletal diseases that could interfere the study.

Study design This was a single-centre, cross-sectional study.

Intervention： Inspiratory resistive training All participants conducted inspiratory resistive training using inspiratory resistive trainer (PFLEX, Respironics Inc, USA). Pdi and EMGdi were recorded synchronously.Inspiratory resistive load was change from low intensity into moderate and high intensity randomly（inspiratory hole diameters was set to 5.3mm, 2.4mm and 1.8mm,respectively）

Inspiratory threshold load training Inspiratory threshold load training was conducted by all participants using the inspiratory threshold load trainer (Threshold Inspiration Muscle Trainer, Respironics Inc, USA) .Inspiratory threshold pressure was set to low, medium and high intensity randomly（threshold pressure was 30%,60% and 80% of MIP, respectively).

Measurements ：transdiaphragmatic pressure and neural respiratory drive

ELIGIBILITY:
Inclusion Criteria:

1. Severe and very severe COPD (postbronchodilator FEV1/FVC under 70% and FEV1 under 50% of the predicted value (GOLD C and D group);
2. Inspiratory muscle weakness（Maximal Inspiratory Pressure under 60cmH2O）;
3. Bronchial dilation test (BDT) negative

Exclusion Criteria:

1. acute exacerbation in the previous 4 weeks;
2. using the oral corticosteroids within 4 weeks;
3. history of other respiratory, cardiovascular, neuromuscular, musculoskeletal diseases that could interfere the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
transdiaphragmatic pressure | half an hour

SECONDARY OUTCOMES:
neural respiratory drive | half an hour

CONTACTS AND LOCATIONS:
Overall Officials: Rongchang Chen, Master, Study Chair — Guangzhou Institude of Respiratory Disease

IPD SHARING:
Plan to Share IPD: Undecided